CLINICAL TRIAL: NCT06233448
Title: Thorathic Fluid Content as an Early Predictor of Weaning From Mechanical Ventilation in Acute Respiratory Distress Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mei K abdallah, MD, Principal investigator, Tanta University
Other Study IDs: 36264PR504/1/24
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-01

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Indirect cardiometry — Measurements of thorathic fluid content

SUMMARY:
Thorathic fluid content measurement using indirect cardiometry is required for prediction of Weaning from mechanical ventilation in cases of acute respiratory distress syndrome and its value in sucsess Weaning

ELIGIBILITY:
Inclusion Criteria:

* patients with ARDS on ventilator for more than 48 hr. proceed for extubation

Exclusion Criteria:

* heart, renal, hepatic failure Obesity , pregnancy Pneumothorax, pneumonia, hemorrhage

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult Patient with ARDS on ventilator in our ICU prepared for weaning
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2024-12-02 (Estimated); Study Completion 2024-12-08 (Estimated)

PRIMARY OUTCOMES:
Success of weaning from mechanical ventilation | 48 hours
  Number of participants without artificial aids for ventilation

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University hospitals, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No